CLINICAL TRIAL: NCT06783192
Title: A Study to Assess the Effects of Single Oral Doses of MK-8527 on the Single-Dose Pharmacokinetics of an Oral Contraceptive (Levonorgestrel and Ethinyl Estradiol) in Healthy Adult Postmenopausal or Oophorectomized Female Subjects
Brief Title: A Drug-Drug Interaction Study of MK 8527 With a Combined Oral Contraceptive (LNG/EE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 8527-006
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Human Immunodeficiency Virus (HIV); HIV Pre-Exposure Prophylaxis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1: All Participants (Experimental): Participants receive single doses of LNG/EE alone and in combination with a single dose of MK-8527.
  Interventions: Drug: MK-8527; Drug: LNG/EE

INTERVENTIONS:
Drug: MK-8527 — MK-8527 capsule taken by mouth
Drug: LNG/EE — LNG/EE combination tablet taken by mouth.
  Other Names: levonorgestrel/ethinyl estradiol

SUMMARY:
This study is designed to assess the effect of a single dose of MK-8527 on the single-dose pharmacokinetics (PK) and the safety and tolerability of levonorgestrel/ethinyl estradiol (LNG/EE) in healthy adult postmenopausal or ovariectomized female participants.

ELIGIBILITY:
Inclusion Criteria:

* is in good overall health
* assigned female at birth

Exclusion Criteria:

* has a history of clinically significant endocrine, GI, cardiovascular, hematological, thromboembolic, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* is mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of clinically significant psychiatric disorder of the last 5 years
* has a history of cancer (malignancy)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 14 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Area under the curve from dosing to infinity (AUC0-∞) of LNG alone and with MK-8527 | Up to ~96 hours postdose
Maximum plasma concentration (Cmax) of LNG alone and with MK-8527 | Up to ~96 hours postdose
Time to Cmax (Tmax) of LNG alone and with MK-8527 | Up to ~96 hours postdose
Apparent half-life (t½) of LNG alone and with MK-8527 | Up to ~96 hours postdose
AUC0-∞ of EE alone and with MK-8527 | Up to ~72 hours postdose
Tmax of EE alone and with MK-8527 | Up to ~72 hours postdose

SECONDARY OUTCOMES:
Percentage of participants with ≥1 adverse event (AE) | Up to ~28 days
Percentage of participants discontinuing from study therapy due to AE | Up to ~28 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- QPS-MRA, LLC-Early Phase (Site 0001), South Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com